CLINICAL TRIAL: NCT01573793
Title: Promoting Optimal Parenting
Brief Title: Promoting Optimal Parenting (Bright Start)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Dimitri Christakis, Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 13852; 1R01HD068478-01A1 (NIH)
Record Dates: First submitted 2012-03-30; First posted 2012-04-10 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Cognitive Development; Emotional Development

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Will receive parenting educational materials hypothesized to enhance emotional and cognitive development
  Interventions: Behavioral: Parenting Education
- Control (Sham Comparator): Will receive safety and dental hygiene materials that have no bearing on emotional and cognitive development
  Interventions: Behavioral: Control Group - Safety Materials

INTERVENTIONS:
Behavioral: Parenting Education — Will receive parenting educational materials hypothesized to enhance emotional and cognitive development
  Arms: Intervention
Behavioral: Control Group - Safety Materials — Will receive safety and dental hygiene materials that have no bearing on emotional and cognitive development
  Arms: Control

SUMMARY:
The purpose of this study is to determine if providing parenting education materials delivered in different ways during the first 30 months of a child's life will increase child-parent attachment and promote mother-child interaction, if certain types of strategies improve cognitive, language, and emotional development in infants and toddlers, and if our way of delivering these materials is cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* 18-23 year-old first-time mother of a healthy newborn

Exclusion Criteria:

* Anything other than above

Ages: 18 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-04; Primary Completion 2016-05 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Language ENvironment Analysis System (LENA) | 6/18/30 months - tracking changes throughout study
Adaptive Behavior Assessment System, Second Edition (ABAS-II) | Month 12/24/36/42 - tracking changes throughout study
Brief Infant Sleep Questionnaire(BISQ) | Month 12/24 - tracking changes throughout study
Behavior Rating Inventory of Executive Function - Preschool Version (BRIEF-P) | Month 24/42 - tracking changes throughout study
MacArthur Communicative Development Inventory- Short Form (CDI) | Month 24/42 - tracking changes throughout study
Children's Sleep Habits Questionnaire (CSHQ) | Month 36/42 - tracking changes throughout study
Devereux Early Childhood Assessment-Clinical Form (DECA-C) | Month 24/36/42 - tracking changes throughout study
Devereux Early Childhood Assessment- Infant/Toddler (DECA-I/T) | Month 12
Family Resource Scale (FRS) | Baseline
MARLOWE-CROWNE | Baseline
Maternal Emotional Styles Questionnaire (MESQ) | Month 36
Patient Health Questionnaire 2 (PHQ-2) | Baseline and Month 12/24/36/42 - tracking changes throughout study
Preschool Language Scale-5 (PLS-5) | Month 36
Parenting Sense of Competence-Efficacy(PSOC) | Baseline and Months 12/24/36/42 - tracking changes throughout study
Social competence subscale of the Social Competence and Behavior Evaluation(SCBE) | Months 36/42 - tracking changes throughout study
(Strange Situation Procedure) SSP | Month 15
Nursing Child Assessment Teaching Scale (NCATS) | Months 15/36 - tracking changes throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri A Christakis, MD, MPH, Principal Investigator — Seattle Children's Research Institute, University of Washington
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States